CLINICAL TRIAL: NCT00115908
Title: A Phase 2b, Randomized, Multi-Center, Active-Controlled, Open-Label Study to Evaluate the Efficacy and Safety of Albuferon (Recombinant Human Albumin-Interferon Alfa Fusion Protein) in Combination With Ribavirin in Interferon Alfa Naive Subjects With Chronic Hepatitis C Genotype 1
Brief Title: A Study of Albuferon and Ribavirin in Interferon Naive Subjects With Chronic Hepatitis C Genotype 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALFR-HC-04
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — albuferon; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Albuferon
Drug: Ribavirin
Drug: PEG-IFNalfa2a

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of Albuferon in combination with ribavirin in interferon (IFN) alfa treatment-naïve subjects with chronic hepatitis C genotype 1. The study will randomize subjects to 1 of 4 treatment groups including 3 different Albuferon groups or to the active control group, peginterferon alfa-2a (PEGASYS, PEG-IFNalfa-2a). All subjects will also receive oral daily ribavirin.

ELIGIBILITY:
Key Inclusion Criteria:

* Interferon treatment naive subjects with chronic hepatitis C, HCV genotype 1.
* Compensated liver disease

Key Exclusion Criteria:

* Pregnant or lactating female or males with a pregnant partner.
* A positive test for serum antibodies to the human immunodeficiency virus (HIV-1) or serum hepatitis B virus surface antigen (HBsAg).
* A history of moderate, severe or uncontrolled psychiatric disease.
* A history of immunologically mediated disease, seizure disorder, chronic cardiac disease, chronic pulmonary disease, hemoglobinopathy, coagulopathy, or malignancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2005-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response (SVR), defined as undetectable HCV RNA at 24 weeks after the end of therapy.

SECONDARY OUTCOMES:
Virologic response at Week 4 (VR4), defined as undetectable HCV RNA or a > 2-log reduction in HCV RNA.
Early virologic response at Week 12 (EVR12), defined as undetectable HCV RNA or a > 2-log reduction in HCV RNA.
Undetectable HCV RNA at Week 24.
End of treatment response (ETR), defined as undetectable HCV RNA at Week 48

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (87):
- Australia (16):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Brisbane Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - St. Vincents Hospital, East Melbourne, Victoria
  - Western Hospital, Footscray, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Canada (12):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of Alberta- Liver Unit, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Dalhousie University, Halifax, Nova Scotia
  - McMaster Clinic - Hamilton General Hospital, Hamilton, Ontario
  - University of Western Ontario, London, Ontario
  - Ottawa Civic Hospital, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - University of Saskatchewan, Saskatoon, Saskatchewan
- Czechia (8):
  - FN Bohunice, Brno
  - Klinika infekcnich nemoci, Hradec Králové
  - Nemocnice s poliklinikou Melnik, Mělník
  - Slezska nemocnice, Opava
  - Vseobecna fakultni nemocnice, Prague
  - Nuselska poliklinika - Remedis, Prague
  - Fakultni Thomayerova nemocnice, Prague
  - Ambulance pro interni a infekcni nemoci, Ústí nad Labem
- France (15):
  - University of Angers, CHU Angers, Angers
  - University of Clichy, Hopital Beaujon, Clichy
  - University of Creteil, Hopital Henri Mondor, Créteil
  - University of Grenoble, Hopital Nord, Grenoble
  - University of Lille, Hopital Claude Huriez, Lille
  - University of Lyon, Hopital de l'Hotel Dieu, Lyon
  - University of Marseille, Hopital Saint Joseph, Marseille
  - University of Nice, Hopital de l'Archet, Nice
  - University of Orleans, Hopital de la Source, Orléans
  - University of Paris, Hopital Saint-Antoine, Paris
  - University of Paris, Hopital Pitie-Salpetriere, Paris
  - University of Paris, Hopital Necker, Paris
  - Hopital Haut-Leveque, Pessac
  - University of Toulouse, Clinique Dieulafoy, Toulouse
  - Hopital de Brabois, Vandœuvre-lès-Nancy
- Germany (14):
  - University of Berlin, Charite Campus Virchow Klinikum, Berlin
  - University of Bochum, Kliniken Bergmannsheil, Bochum
  - University of Duesseldorf, Düsseldorf
  - University of Essen, Essen
  - University of Frankfurt, Frankfurt
  - University of Freiburg, Freiburg im Breisgau
  - University of Hamburg, Hospital Hamburg Eppendorf, Hamburg
  - University of Hannover, Hanover
  - University of Heidelberg, Heidelberg
  - University of Saarland, Homburg
  - University of Kiel, Kiel
  - University of Leipzig, Leipzig
  - University of Mainz, Mainz
  - University of Tuebingen, Tübingen
- Israel (6):
  - B´nai-Zion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Hadassah Medical Organization, Jerusalem
  - Holy Family Hospital, Nazareth
  - Rabin Medical Center, Beilinson Campus, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Poland (11):
  - Oddzial Chorob Watroby, Bialystok
  - Katedra i Klinika Chorob Zakaznych i Hepatologii, Bydgoszcz
  - Katedra i Oddzial Kliniczny Chorob Zakaznych, Chorzów
  - Wojewodzki Szpital Zespolony, Kielce
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Klinika Obserwacyjno Zakazna, Lodz
  - Oddzial Zakazny, Poznan
  - Katedra i Klinika Chorob Zakaznych, Szczecin
  - I Oddzial Dzienny SPZOZ, Warsaw
  - Klinika Hepatologii i Nabytych Niedoborow Immunologicznych, Warsaw
  - Katedra i Klinika Chorob Zakaznych, Wroclaw
- Romania (5):
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul de Boli Infectioase si Tropicale "Dr. Victor Babes", Bucharest
  - Spitalul Clinic de Adulti Cluj-Napoca, Cluj-Napoca
  - Institutul de Gastroenterologie si Hepatologie, Iași

REFERENCES:
- [Derived] Neumann AU, Pianko S, Zeuzem S, Yoshida EM, Benhamou Y, Mishan M, McHutchison JG, Pulkstenis E, Mani Subramanian G. Positive and negative prediction of sustained virologic response at weeks 2 and 4 of treatment with albinterferon alfa-2b or peginterferon alfa-2a in treatment-naive patients with genotype 1, chronic hepatitis C. J Hepatol. 2009 Jul;51(1):21-8. doi: 10.1016/j.jhep.2009.01.017. Epub 2009 Mar 11. PMID 19447518
- [Derived] Zeuzem S, Yoshida EM, Benhamou Y, Pianko S, Bain VG, Shouval D, Flisiak R, Rehak V, Grigorescu M, Kaita K, Cronin PW, Pulkstenis E, Subramanian GM, McHutchison JG. Albinterferon alfa-2b dosed every two or four weeks in interferon-naive patients with genotype 1 chronic hepatitis C. Hepatology. 2008 Aug;48(2):407-17. doi: 10.1002/hep.22403. PMID 18666223